CLINICAL TRIAL: NCT00028873
Title: An EORTC-IDBBC/ECSG Phase II Study Evaluating The Role Of The Multi-Drug Resistance (MDR) Reversor, R101933, In Patients With Taxane Refractory Metastatic Breast Cancer
Brief Title: R101933 Combined With Chemotherapy in Treating Patients With Metastatic Breast Cancer That Has Not Responded to Previous Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-10003-16004; EORTC-16004; ECSG-EORTC-16004; IDBBC-10003
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; laniquidar; Paclitaxel

INTERVENTIONS:
Drug: docetaxel
Drug: laniquidar
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Some tumors become resistant to chemotherapy drugs. Combining R101933 with paclitaxel or docetaxel may reduce resistance to the drug and allow the tumor cells to be killed.

PURPOSE: Phase II trial to study the effectiveness of combining R101933 with either paclitaxel or docetaxel in treating patients who have metastatic breast cancer that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the activity of R101933 in combination with paclitaxel or docetaxel in terms of response to treatment and level of clinical benefit in patients with taxane-refractory metastatic breast cancer.
* Determine the safety of this regimen in these patients.
* Determine the acute side effects in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive R101933 IV over 1 hour immediately followed by paclitaxel IV over 3 hours or docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for 7 courses in the absence of disease progression or unacceptable toxicity. Patients who have no disease progression after 7 courses may continue with treatment at the investigator's discretion.

Patients are followed every 6 weeks until disease progression.

PROJECTED ACCRUAL: A total of 12-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic breast cancer
* Received at least 2 prior courses of paclitaxel-based chemotherapy at doses between 175-200 mg/m^2 (given over 3 hours every 3 weeks) or docetaxel-based chemotherapy at doses between 75-100 mg/m^2 (given over 1 hour every 3 weeks) as most recent anticancer therapy
* Evidence of disease resistance

  * Progressive disease as best response OR
  * Transient response or disease stabilization followed by progression during taxane-based treatment
  * Disease progression on a combination of a taxane and another cytotoxic agent allowed
* Unidimensionally measurable disease

  * At least 1 target lesion that clearly progressed or developed during prior taxane therapy
  * Lesions stable or responsive to prior taxane therapy are not considered target lesions
  * Lesions that have been irradiated within the past 3 months are not considered target lesions unless they have clearly progressed or appeared since radiotherapy
* No bone metastases as only site of measurable disease
* No rapidly progressive visceral metastases
* No symptomatic CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Not specified

Menopausal status:

* Not specified

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Transaminases no greater than 2.5 times ULN (5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 1.5 times ULN
* Calcium normal

Cardiovascular:

* LVEF normal by echocardiogram (ECG) or MUGA scan
* QTc less than 450 sec on baseline ECG
* No prior clinically significant arrhythmias requiring treatment
* No cardiac infarction
* No atrial ventricular enlargement or hypertrophy

Other:

* No prior toxicity to paclitaxel that would preclude study dose and schedule
* Sodium, potassium, chloride, and bicarbonate normal
* No pre-existing neuropathy greater than grade 2
* No other prior or concurrent malignancy except adequately treated carcinoma in situ of the cervix, contralateral breast cancer, or nonmelanoma skin cancer or cancer that has been in remission for more than 5 years
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent anticancer biologic agents

Chemotherapy:

* See Disease Characteristics
* No more than 8 weeks since last course of prior taxane-based chemotherapy
* No more than 2 prior chemotherapy regimens for metastatic breast cancer
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* No concurrent anticancer hormonal therapy

Radiotherapy:

* See Disease Characteristics
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No prior multi-drug resistance inhibitor
* No new anticancer therapy initiation since last course of prior taxane-based chemotherapy
* No concurrent angiotensin converting enzyme inhibitor and/or drugs that may prolong the QTc interval
* No other concurrent anticancer therapy
* Concurrent bisphosphonates for treatment and prevention of bony metastases allowed provided drugs were initiated prior to study (treatment of hypercalcemia due to malignancy allowed regardless of time of initiation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2001-09; Primary Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo L. Rapoport, MD, MMed(IntMed), Study Chair — Medical Oncology Centre of Rosebank; Pierre Fumoleau, MD, PhD, Study Chair — Centre Georges Francois Leclerc; Martine J. Piccart-Gebhart, MD, PhD, Study Chair — Jules Bordet Institute
Locations (2):
- Institut Jules Bordet, Brussels, Belgium
- CRLCC Nantes - Atlantique, Nantes-Saint Herblain, France